CLINICAL TRIAL: NCT05778747
Title: Feasibility of the Heart to Heart Yoga Program in Patients With Heart Failure and Caregivers
Brief Title: Feasibility of the Heart to Heart Yoga Program
Acronym: H2HYoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misook L. Chung (Other)
Responsible Party: Sponsor-Investigator, Misook L. Chung, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 72684
Record Dates: First submitted 2022-06-22; First posted 2023-03-21 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure; Caregiver Burden; Depression; Anxiety; Stress
Keywords: Caregiver; Yoga
MeSH Terms: conditions — Heart Failure; Caregiver Burden; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A total of 20 patients with HF and 20 caregivers (n= 40) who have at least mild depressive symptoms (Patient Health Questionnaire 9 [PHQ-9] score = 5) will be randomly assigned to the intervention or usual care group stratified by patient and caregiver groups (Figure 1). Only participants in the intervention will be asked to attend the 12-week sessions (two sessions per week; a total of 24 sessions in 12 weeks) via video conferencing (i.e., ZOOM). The short-term intervention efficacy will be assessed at the following week of the completion of 12-weeks sessions. Primary psychological outcomes include depressive symptoms, anxiety, stress, and quality of life. Primary physical outcomes include physical activity level, sleep quality, and perceived symptoms.
  Interventions: Other: Heart to Heart Yoga
- Usual Care (No Intervention): Participants in the usual care group will also receive the printed information and links to the AHA's Life's Simple 7 program without explicit skills and training, including education and stress management. We will encourage stress management by watching and practicing yoga programs by providing a yoga mat.

INTERVENTIONS:
Other: Heart to Heart Yoga — The Heart to Heart Yoga intervention is a therapeutic and standardized form of yoga intervention that is adapted from MediYoga designed to fit the needs of patients with HF and family caregivers who have physical limitations and depressive symptoms and to fit cultural and social norms in Kentucky. The intervention will use a gradual, physical/ psychological yoga adaptation approach, and it will be delivered two times per week (40 -60 minutes per session) via videoconference technology for 12 weeks (total 24 sessions). Real-time, face-to-face, video conferencing technology is used.
  Arms: Intervention

SUMMARY:
A two-group (intervention vs. usual care), randomized controlled design will be used to determine the feasibility and acceptability of the intervention, the Heart2Heart program, and determine efficacy on physical and psychological outcomes in patients with heart failure (HF) and caregivers. A total of 20 patients with HF and 20 caregivers (n= 40) will be randomly assigned to the intervention or usual care group stratified by patient and caregiver groups. Only participants in the intervention will be asked to attend the 12-week sessions (two sessions per week; a total of 24 sessions in 12 weeks) via video conferencing (i.e., ZOOM). The short-term intervention efficacy will be assessed following week of the completion of 12-weeks sessions. Primary psychological outcomes include depressive symptoms, anxiety, stress, and quality of life. Primary physical outcomes include physical activity level, sleep quality, and perceived symptoms.

DETAILED DESCRIPTION:
Heart2Heart Intervention. In this study, the Heart to Heart Yoga intervention is a therapeutic and standardized form of yoga intervention that is adapted from MediYoga designed to fit the needs of patients with heart failure (HF) and family caregivers who may have physical limitations and to fit cultural and social norms in Kentucky. The Heart to Heart Yoga intervention key personnel include two primary investigators, two professional yoga instructors, and one PhD student who are all nurses and were certified Medi-Yoga instructor Level 1 by completing more than 120 hours of Medi-yoga training course for medical professionals. The intervention will use a gradual, physical/ psychological yoga adaptation approach, and it will be delivered two times per week (40 -60 minutes per session) via videoconference technology for 12 weeks (total 24 sessions). Real-time, face-to-face, video conferencing technology is used. In the recent systematic literature review, yoga has been delivered for 12 weeks in patients with HF. The the12-week duration was selected in this study by considering variations of individual adaptation and available evidence in the literature. Yoga sessions will be delivered by two registered nurses who were yoga instructors and certified MediYoga instructors.

The 12-weeks of intervention include three structured sessions. At each session, the first part will focus on deep breathing (5- 11 minutes), followed by physical posture movement (3 -11 minutes), and then meditation (6 -11 minutes), based on the structured gradual adaptation program. Participants will be instructed to modify movements to ensure comfort and safety. For example, if a participant is more comfortable seated in a chair instead of the floor, the instructor will demonstrate exercise modification while ensuring target muscles are utilized. All sessions will be delivered as group sessions using a video-conferencing program on a digital multimedia device. Each week, three yoga sessions are available to allow participants flexibility in attendance. The intervention group also receives a short-video clip each week (up to 10 minutes) and recommend to follow to practice yoga for 10 minutes per day, and a total of 50 minutes per week while not attending sessions. Participants will record practice time in a Yoga log booklet.

The investigators will limit the number of participants up to 10 at each session by monitoring enrollment rates. Participants will also receive materials that include yoga poses guides and mats. Without explicit skill demonstration and training, the intervention group will receive the printed information and links to the AHA's Life's Simple 7 program.

Usual Care Group. Participants in the usual care group will also receive the printed information and links to the AHA's Life's Simple 7 program without explicit skills and training, including education and stress management. Stress management will be encouraged by watching and practicing yoga programs by providing a yoga mat.

ELIGIBILITY:
Inclusion Criteria Patients:

* diagnosis of chronic HF confirmed by their cardiologist with either preserved or reduced ejection fraction
* be able to speak and write English.

Inclusion Criteria Caregivers:

* be a primary caregiver identified by the patient
* the spouse, committed partner, or family member living with the HF patient
* be able to speak and understand English
* ability to give informed consent
* have no major comorbidities (i.e., HF, and terminal illness including active cancer, renal/liver failure) to perform yoga practice.

Exclusion Criteria:

* After obtaining the signed consent, we will screen depressive symptoms using the 9-items of the Patient Health Questionnaire (see the detailed process of screening depressive symptom criterion in the procedure) because we will target only patients and caregivers who experience at least mild depressive symptoms.
* major clinical cognitive impairment (i.e., dementia, Alzheimer's disease, and severe stroke)
* co-existing terminal illness (e.g., cancer)
* major psychiatric disorder other than depression
* referral for heart transplantation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Feasibility of Intervention | 12 weeks
  Intervention evaluations will include a Likert style questionnaire to assess feasibility.
  Open-ended questions and comments will be utilized to gather additional information on any barriers or facilitators of participation and completion. feasibility data will be collected by each group's recruitment and retention rates by tracking eligible and enrolled participants using the consort diagram. We will also track participants' attendance rates and total attendance time (minutes) by monitoring the recorded sessions for the intervention acceptability. We will also collect participants' intervention satisfaction, enjoyment of the session, willingness to engage in yoga at home, and difficulty following yoga instruction using an 11-point numeric analog scale (0= not at all,10= very much) each session. We will also collect the Treatment Acceptability Adherence Scale (TAAS) and the Client Satisfaction Questionnaire (CSQ).
Physical activity | 12 weeks
  Sit and stand
Physical activity | 12 weeks
  Activity energy expenditure using accelerometer of activity monitor device (ActiGraph)
Sleep Quality | 12 weeks
  Pittsburgh Sleep Quality Index
Sleep Quality | 12 weeks
  Actigraphy data
C Reactive Protein | 12 weeks
Interleukin 6 | 12 weeks
Brain Derived Neurotrophic Factor | 12 weeks
Perceived Symptoms | 12 weeks
  Heart Failure Somatic Symptom Checklist
Perceived Symptoms | 12 weeks
  Memorial Symptoms Assessment Scale
Depressive Symptoms | 12 weeks
  Patient Health Questionnaire-9 (PHQ-9)
Anxiety | 12 weeks
  Hospital Anxiety and Depressive Symptoms Scale (HADS)
Stress | 12 weeks
  Cohen's Perceived Stress Scale
Stress | 12 weeks
  Salivary cortisol awakening response
Caregiver Burden | 12 weeks
  Zarit Burden Interview (ZBI)
Caregiver Burden | 12 weeks
  Oberst Caregiving Burden Scale (OCBS)
Caregiver Burden | 12 weeks
  Caregiving Burden Questionnaire for heart failure (CBQ-HF)
Quality of Life | 12 weeks
  European Quality of Life (EQ-5D)
Quality of Life | 12 weeks
  Minnesota Living with Heart failure (MLHFQ)

CONTACTS AND LOCATIONS:
Overall Officials: Misook Chung, PhD, RN, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No